CLINICAL TRIAL: NCT01605214
Title: Measurement of Extravascular Lung Water to Detect and Predict Primary Graft Dysfunction Following Lung Transplant
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Toronto General Hospital (Other)
Responsible Party: Principal Investigator, John Granton, Dr. John T. Granton, Professor, Division Head of Respirology, University Health Network, Toronto
Other Study IDs: UHNEVLW-1
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Primary Graft Dysfunction
Keywords: Extravascular Lung Water; Transpulmonary Thermodilution; Primary Graft Dysfunction; Ischemia Reperfusion Injury
MeSH Terms: conditions — Primary Graft Dysfunction; Reperfusion Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bilateral Lung Transplant: All patients undergoing bilateral lung transplant for any indication will be considered for enrollment in the study. The characteristics of measurements of extravascular lung water will be compared following surgery in those who develop primary graft dysfunction compared to those who do not.

SUMMARY:
Primary graft dysfunction (PGD) is the most common cause of early morbidity and mortality following lung transplant and is characterized by acute lung injury and capillary leak leading to an increase in extravascular lung water index (ELWI) and impaired graft function. PGD has many features in common with acute respiratory distress syndrome (ARDS). PGD may be life-threatening and can also lead to impaired long term lung function. In ARDS, a restrictive fluid strategy has been associated with an improvement in lung function and outcomes. Accurate methods of evaluating, quantifying and guiding the hemodynamic / fluid management and limiting the extent of ELWI that accumulates in the setting of PGD are lacking. Using transpulmonary thermodilution to estimate ELWI and the pulmonary permeability index (PPI) represents a novel approach to fluid management, which has been used in patients with ARDS, but to date not in the transplant setting. To determine if these measurements may better guide the management of lung transplant patients, the investigators first wish to establish whether these methods are able to predict the onset of clinical pulmonary edema earlier, whether they correlated with traditional markers of PGD, and whether they may be useful for predicting outcomes.

AIM 1: The investigators will evaluate the correlation between ELWI and current surrogates of pulmonary edema in lung transplant patients with and without Primary Graft Dysfunction (PGD)

AIM 2: The investigators will correlate the use of ELWI and PPI to determine the presence and severity of PGD.

AIM 3: a) The investigators will determine whether early measurements of ELWI and PPI can predict the onset of PGD.

b) Across different strata of PGD, the investigators will determine whether ELWI and PPI have a differential effect on duration of mechanical ventilation.

The results of the study will be used for the following:

1. Provide the rationale for routine monitoring of ELWI to detect PGD if found to be more discriminatory and have a stronger association with outcome compared to the current gold standard.
2. Provide the means of early identification of those as risk of developing PGD in order to guide management decisions or future therapeutic interventions aimed at preventing or treating PGD.
3. Provide the requisite groundwork for a clinical trial comparing the effects of an ELWI-driven protocol versus usual care on ICU outcomes in lung transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive bilateral lung transplant recipients

Exclusion Criteria:

* Immediate need for extracorporeal life support following transplant (those requiring ECLS four hours after intensive care admission can be included as the investigators would have obtained some ELWI measurements)
* Contraindications to femoral artery catheterization (eg, abdominal aortic aneurysm)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing bilateral lung transplant for any indication will be considered to be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
AIM 1: The presence of pulmonary edema on chest X ray (CXR) at 24 hours determined by blinded CXR reviewers | 24 hours following lung transplant
  On post operative day 1 (24 hours following lung transplant), the investigators will evaluate whether extravascular lung water measured at 24 hours correlates with pulmonary edema determined by reviewers of the CXR blinded to the extravascular lung water measurement. The investigators will use Pearson's correlation for normally distributed and Spearman's correlation for non-normally distributed values. A correlation coefficient of >0.8 will be considered a strong correlation
AIM 2: The presence of primary graft dysfunction at 24 hours determined by CXR evidence of bilateral airspace disease and Pa02/FiO2 ratio threshold by reviewers blinded to the extravascular lung water and pulmonary permeability measurements at 24 | 24 hours
  24 hours following lung transplant, the investigators will evaluate whether the combination of extravascular lung water and pulmonary permeability measurements at 24 hours correlate with the presence and severity of primary graft dysfunction (PGD) at 24 hours. The median extravascular lung water and pulmonary permeability measurements will be calculated. The combinations of above/below median extravascular lung water with above/below median pulmonary permeability will be correlated to the presence of PGD. (eg. high ELWI + high PPI, high ELWI + low PPI, low ELWI + high PPI, low ELWI + low PPI) using Pearson's and Spearman's correlation where appropriate.
  Grade 0 PGD - Normal CXR AND a PaO2/FiO2 >300mmHg Grade 1 PGD - Bilateral airspace disease on CXR with AND a PaO2/FiO2 >300mmHg Grade 2 PGD - Bilateral airspace disease on CXR with AND a PaO2/FiO2 200-300mmHg Grade 3 PGD - Bilateral airspace disease on CXR with AND a PaO2/FiO2 <200mmHg.
AIM 3: The presence of primary graft dysfunction at 24 hours determined by CXR and Pa02/FiO2 ratio by reviewers blinded to early (time 0) extravascular lung water and pulmonary permeability measurements | Time 0 extravascular lung water and pulmonary permeability measurements and primary graft dysfunction at 24 hours
  The investigators will compare whether immediate (time 0) post operative measurements of the combination of extravascular lung water and pulmonary permeability can predict the later onset (24 hours) of primary graft dysfunction. The combinations of above/below median extravascular lung water with above/below median pulmonary permeability will be correlated to the presence of PGD. (eg. high ELWI + high PPI, high ELWI + low PPI, low ELWI + high PPI, low ELWI + low PPI) using logistic regression.
  Grade 0 PGD - Normal CXR AND a PaO2/FiO2 >300mmHg Grade 1 PGD - Bilateral airspace disease on CXR with AND a PaO2/FiO2 >300mmHg Grade 2 PGD - Bilateral airspace disease on CXR with AND a PaO2/FiO2 200-300mmHg Grade 3 PGD - Bilateral airspace disease on CXR with AND a PaO2/FiO2 <200mmHg.

SECONDARY OUTCOMES:
AIM 1: The presence of pulmonary edema on chest X ray at 48 and 72 hours evaluated by CXR reviewers blinded to the extravascular lung water measurements measured at 48 and 72 hours | 48 and 72 hours following lung transplant
  On post operative day 2 and 3 (48 and 72 hours following lung transplant), the investigators will evaluate whether the extravascular lung water measurements taken at 48 and 72 hours correlate with pulmonary edema determined by CXR. The investigators will use Pearson's correlation for normally distributed and Spearman's correlation for non-normally distributed values. A correlation coefficient of >0.8 will be considered a strong correlation
AIM 2: The presence of late primary graft dysfunction determined by CXR and PaO2/FiO2 ratio evaluated by reviewers blinded to the extravascular lung water and pulmonary permeability measurements evaluated at 48 and 72 hours | 48 and 72 hours following lung transplant
  On post operative day 2 and 3 (48 and 72 hours following lung transplant), the investigators will evaluate whether the combination of of extravascular lung water and pulmonary permeability measurements taken at 48 and 72 hours correlate with the presence and severity of primary graft dysfunction (PGD). The combinations of above/below median extravascular lung water with above/below median pulmonary permeability will be correlated to the presence of PGD. (eg. high ELWI + high PPI, high ELWI + low PPI, low ELWI + high PPI, low ELWI + low PPI) using Pearson's and Spearman's correlation where appropriate.
  Grade 0 PGD - Normal CXR AND a PaO2/FiO2 >300mmHg Grade 1 PGD - Bilateral airspace disease on CXR with AND a PaO2/FiO2 >300mmHg Grade 2 PGD - Bilateral airspace disease on CXR with AND a PaO2/FiO2 200-300mmHg Grade 3 PGD - Bilateral airspace disease on CXR with AND a PaO2/FiO2 <200mmHg.
AIM 3: The presence of late primary graft dysfunction (48 and 72 hours) determined by CXR and PaO2/FiO2 ratio evaluated by reviewers blinded to the extravascular lung water and pulmonary permeability measurements at time 0 | Extravascular lung water and pulmonary permeability measurements at time 0 hours, primary graft dysfunction determination at 48 or 72 hours
  The investigators will evaluate whether the early (time 0 hours) measurements of the combination of extravascular lung water and pulmonary permeability index can predict the development of late primary graft dysfunction (PGD) at 48 hours or 72 hours. The combinations of above/below median extravascular lung water with above/below median pulmonary permeability will be correlated to the presence of PGD. (eg. high ELWI + high PPI, high ELWI + low PPI, low ELWI + high PPI, low ELWI + low PPI) using Pearson's and Spearman's correlation where appropriate.
  Grade 0 PGD - Normal CXR AND a PaO2/FiO2 >300mmHg Grade 1 PGD - Bilateral airspace disease on CXR with AND a PaO2/FiO2 >300mmHg Grade 2 PGD - Bilateral airspace disease on CXR with AND a PaO2/FiO2 200-300mmHg Grade 3 PGD - Bilateral airspace disease on CXR with AND a PaO2/FiO2 <200mmHg.
AIM 3: The presence of any primary graft dysfunction determined by CXR and PaO2/FiO2 ratio (24, 48 or 72 hours) evaluated by reviewers blinded to the early extravascular lung water and pulmonary permeability measurements (6 hours and 12 hours) | Extravascular lung water and pulmonary permeability measurements at 6 hours and 12 hours, any primary graft dysfunction determined at 24, 48 or 72 hours
  The investigators will evaluate whether the early (time 6 hours and 12 hours) measurements of the combination of extravascular lung water and pulmonary permeability index can predict the development of primary graft dysfunction (PGD) at 24, 48 or 72 hours. The combinations of above/below median extravascular lung water with above/below median pulmonary permeability will be correlated to the presence of PGD. (eg. high ELWI + high PPI, high ELWI + low PPI, low ELWI + high PPI, low ELWI + low PPI) using logistic regression.
  Grade 0 PGD - Normal CXR AND a PaO2/FiO2 >300mmHg Grade 1 PGD - Bilateral airspace disease on CXR with AND a PaO2/FiO2 >300mmHg Grade 2 PGD - Bilateral airspace disease on CXR with AND a PaO2/FiO2 200-300mmHg Grade 3 PGD - Bilateral airspace disease on CXR with AND a PaO2/FiO2 <200mmHg.
AIM 3: Duration of mechanical ventilation | Extravascular lung water and pulmonary permeability measurements at 24 hours, Hospital admission following lung transplant
  The investigators will evaluate whether extravascular lung water and pulmonary permeability measurements at 24 hours, regardless of primary graft dysfunction grade, correlates with duration of mechanical ventilation during the first intensive care unit stay following lung transplant using linear regression analysis

CONTACTS AND LOCATIONS:
Overall Officials: John Granton, MD, FRCPC, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Monnet X, Anguel N, Osman D, Hamzaoui O, Richard C, Teboul JL. Assessing pulmonary permeability by transpulmonary thermodilution allows differentiation of hydrostatic pulmonary edema from ALI/ARDS. Intensive Care Med. 2007 Mar;33(3):448-53. doi: 10.1007/s00134-006-0498-6. Epub 2007 Jan 13. PMID 17221189
- [Background] Sakka SG, Ruhl CC, Pfeiffer UJ, Beale R, McLuckie A, Reinhart K, Meier-Hellmann A. Assessment of cardiac preload and extravascular lung water by single transpulmonary thermodilution. Intensive Care Med. 2000 Feb;26(2):180-7. doi: 10.1007/s001340050043. PMID 10784306
- [Background] Chung FT, Lin HC, Kuo CH, Yu CT, Chou CL, Lee KY, Kuo HP, Lin SM. Extravascular lung water correlates multiorgan dysfunction syndrome and mortality in sepsis. PLoS One. 2010 Dec 16;5(12):e15265. doi: 10.1371/journal.pone.0015265. PMID 21187890
- [Background] Della Rocca G, Costa GM, Coccia C, Pompei L, Di Marco P, Pietropaoli P. Preload index: pulmonary artery occlusion pressure versus intrathoracic blood volume monitoring during lung transplantation. Anesth Analg. 2002 Oct;95(4):835-43, table of contents. doi: 10.1097/00000539-200210000-00009. PMID 12351254
- [Background] Michard F, Alaya S, Zarka V, Bahloul M, Richard C, Teboul JL. Global end-diastolic volume as an indicator of cardiac preload in patients with septic shock. Chest. 2003 Nov;124(5):1900-8. doi: 10.1378/chest.124.5.1900. PMID 14605066
- [Background] Sakka SG, Klein M, Reinhart K, Meier-Hellmann A. Prognostic value of extravascular lung water in critically ill patients. Chest. 2002 Dec;122(6):2080-6. doi: 10.1378/chest.122.6.2080. PMID 12475851
- [Background] Hillinger S, Hoerstrup SP, Zollinger A, Weder W, Schmid RA, Stammberger U. A new model for the assessment of lung allograft ischemia/reperfusion injury. J Invest Surg. 2000 Jan-Feb;13(1):59-65. doi: 10.1080/089419300272267. PMID 10741952
- [Background] Rocca GD, Coccia C, Costa GM, Pompei L, Di Marco P, Pierconti F, Cappa M, Venuta F, Pietropaoli P. Is very early extubation after lung transplantation feasible? J Cardiothorac Vasc Anesth. 2003 Feb;17(1):29-35. doi: 10.1053/jcan.2003.6. PMID 12635057